CLINICAL TRIAL: NCT05953246
Title: Comparing Designs for Environmental Sustainability "Eco-Labels" for Restaurant Menus
Brief Title: Comparing Designs for Restaurant "Eco-Labels"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Harvard Pilgrim Health Care (Other)
Responsible Party: Principal Investigator, Anna Grummon, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69580b
Record Dates: First submitted 2023-07-11; First posted 2023-07-20 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Food Preferences
Keywords: food labeling; sustainability; diet; food choices
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Neutral labels (Active Comparator): Labels shown will be QR codes with and without neutral text (i.e., not mentioning environmental impacts)
  Interventions: Behavioral: Neutral labels
- Numeric text-only sustainability labels (Experimental): Labels shown will contain numeric text depicting the greenhouse gas emissions associated with production of the menu item
  Interventions: Behavioral: Numeric text-only sustainability labels
- Endorsement text-only sustainability labels (Experimental): Labels shown will contain text endorsing menu items as having low environmental impact
  Interventions: Behavioral: Endorsement text-only sustainability labels
- Endorsement icon-only sustainability labels (Experimental): Labels shown will contain icons endorsing menu items as having low environmental impact
  Interventions: Behavioral: Endorsement icon-only sustainability labels
- Endorsement text-plus-icon sustainability labels (Experimental): Labels shown will contain both text and icons endorsing menu items as having low environmental impact
  Interventions: Behavioral: Endorsement text-plus-icon sustainability labels

INTERVENTIONS:
Behavioral: Neutral labels — Participants view neutral labels (QR codes with and without neutral text) for menu items
  Arms: Neutral labels
Behavioral: Numeric text-only sustainability labels — Participants view labels with numeric text depicting the greenhouse gas emissions associated with production of the menu item
  Arms: Numeric text-only sustainability labels
Behavioral: Endorsement text-only sustainability labels — Participants view labels using text to endorse menu items as having low environmental impact
  Arms: Endorsement text-only sustainability labels
Behavioral: Endorsement icon-only sustainability labels — Participants view labels using icons to endorse menu items as having low environmental impact
  Arms: Endorsement icon-only sustainability labels
Behavioral: Endorsement text-plus-icon sustainability labels — Participants view labels using text and icons to endorse menu items as having low environmental impact
  Arms: Endorsement text-plus-icon sustainability labels

SUMMARY:
The aim of this study is to compare responses to 5 different types of labels for restaurant menus: 1) Control (non-sustainability-label: neutral labels not referencing environmental sustainability); 2) Numeric text-only sustainability label; 3) Endorsement text-only sustainability label; 4) Endorsement icon-only sustainability label; 5) Endorsement text-plus-icon sustainability label. Participants will be randomized to 1 of the 5 labeling arms above. Each participant will view 3 labels (shown in random order) from their randomly assigned labeling arm and respond to survey questions about each label (e.g., attention, perceived effectiveness).

DETAILED DESCRIPTION:
This is an online randomized controlled trial. Investigators will recruit participants through a survey company to complete an online survey. In the study, participants will be randomized to 1 of 5 labeling arms: 1) Control (non-sustainability-label: neutral labels not referencing environmental sustainability); 2) Numeric text-only sustainability label; 3) Endorsement text-only sustainability label; 4) Endorsement icon-only sustainability label; 5) Endorsement text-plus-icon sustainability label. Participants will be randomized to 1 of the 5 labeling arms above. Each participant will view 3 labels (shown in random order) from their randomly assigned labeling arm and respond to survey questions about each label (e.g., attention, perceived effectiveness).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be US adults
* Ages 18 or older
* With an over-sample of adults (50% of total sample) 18-29 years

Exclusion Criteria:

* Younger than 18
* Non-US

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2207 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Perceived message effectiveness | The survey will take up to 20 minutes
  Participants will rate the extent to which the label makes them want to choose items with the label on a 5-point scale ranging from low (1) to high (5). They will also rate the extent to which the label makes eating items with the label seem appealing to them on a 5-point scale ranging from low (1) to high (5). These items are adapted from the 3-item UNC Perceived Message Effectiveness scale. Investigators will average responses to these two items to create a perceived message effectiveness score, which will also range from low (1) to high (5). Higher scores therefore indicate higher perceived message effectiveness.

SECONDARY OUTCOMES:
Attention | The survey will take up to 20 minutes
  Participants will rate the extent to which the label captures their attention on a 5-point response scale ranging from low (1) to high (5). Higher scores indicate more attention-grabbing labels (a better outcome).
Thinking about environmental effects | The survey will take up to 20 minutes
  Participants will rate the extent to which the label makes them think about the environmental impacts of their food choices on a 5-point response scale ranging from low (1) to high (5). Higher scores indicate labels elicit more thinking about environmental effects (a better outcome).
Anticipated social interactions | The survey will take up to 20 minutes
  Participants will rate how likely they are to talk about the label with others in the next week on a 5-point response scale ranging from low (1) to high (5). Higher scores indicate labels elicit more anticipated social interactions (a better outcome).
Believability | The survey will take up to 20 minutes
  Participants will rate how believable the label is on a 5-point response scale ranging from low (1) to high (5). Higher scores indicate labels are more believable (a better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Anna H Grummon, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Stanford School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
In the consenting process, participants agreed that de-identified data produced from this project may be distributed for future research studies without additional informed consent. After analysis, we will upload the de-identified data to ResearchBox for public sharing.
Supporting Information: SAP
Time Frame: Starting 6 months after publication
Access Criteria: Public
URL: https://researchbox.org/